CLINICAL TRIAL: NCT02679248
Title: A Double Blind, Placebo Controlled Parallel Study to Investigate the Effect of a Nitric Oxide Supplementation Product on Pre- and Mildly Hypertensive Adults.
Brief Title: A Study to Investigate the Effect of a Nitric Oxide Supplementation on Pre- and Mildly Hypertensive Adults
Acronym: 15NBHN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: KGK Science Inc. (Industry)
Collaborators: Neogenis Laboratories (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 15NBHN
Record Dates: First submitted 2016-02-03; First posted 2016-02-10 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Pre-hypertension
Keywords: Pre-hypertension; Mild hypertension; Dietary supplement; Efficacy; Nitric oxide; Neo40 Daily
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neo40 Daily® (Experimental)
  Interventions: Dietary Supplement: Neo40 Daily®
- Placebo (Experimental)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Neo40 Daily®
  Arms: Neo40 Daily®
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This study will investigate the effect of a nitric oxide supplementation product, Neo40 Daily®, on blood pressure in pre-hypertensive and mildly hypertensive adults. Subjects will take 2 lozenges per day 12 hours apart for 8 weeks. Half of the subjects will receive Neo40 Daily® and the other half of the subjects will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* If female, subject is not of child bearing potential, which is defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) OR Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:

  * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
  * Double-barrier method
  * Non-hormonal intrauterine devices
  * Vasectomy of partner
* BMI 18.5-29.9 kg/m2 (±1 kg/m2)
* Seated resting systolic blood pressures between 130-150 mmHg (inclusive) and diastolic blood pressure ≤ 100 mmHg at screening visit
* Agreement to maintain current level of physical activity and diet throughout the study
* Agrees to comply with study procedures including willingness to fast at least 12 hours before blood samples, abstain from alcohol two days prior to blood sampling and blood pressure measurement, abstain from coffee at least 14 hours before blood pressure measurement and abstain from physical exercise at least 4 hours before and during blood pressure measurement
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Has given voluntary, written, informed consent to participate in the study
* Use of medication for the treatment of hypertension
* Use of prescription diuretics
* Use of natural health products for the treatment of hypertension within 2 weeks of screening (e.g. garlic supplements, french lavender supplements, cardamom supplements, cinnamon supplements, basil supplements, hawthorn cats claw and celery seed supplements)
* Significant cardiac history defined as a history of myocardial infarction (MI); coronary angioplasty or bypass graft(s); Valvular disease or repair; unstable angina pectoris; transient ischemic attack (TIA); cerebrovascular accidents (CVA); congestive heart failure; coronary artery disease (CAD); or angina (stable or unstable)
* Type I or Type II diabetes
* Diagnosis of hypertensive retinopathy, left ventricular dysfunction or peripheral artery disease
* Abnormal electrolytes, liver or kidney function
* Diagnosis of secondary hypertension
* Diagnosis of anemia
* Unstable medical conditions that in the opinion of the Qualified Investigator preclude the volunteer from participating in the study
* Alcohol or drug abuse within the last 6 months
* Use of medicinal marijuana
* Clinically significant abnormal laboratory results at screening
* Participation in a clinical research trial within 30 days prior to randomization
* Allergy or sensitivity to study supplement ingredients
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2017-02-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Daytime Systolic BP | 8 weeks
  Mean ambulatory BP measured from 8am to 8pm

SECONDARY OUTCOMES:
Daytime Diastolic BP | 8 weeks
  Mean ambulatory BP measured from 8am to 8pm
24-hour BP | 8 weeks
  Measured with ambulatory BP
Night-time BP | 8 weeks
  Mean ambulatory BP measured from 12am to 6am
BP Variability | 8 weeks
  Measured with ambulatory BP
Seated BP | 8 weeks
  Seated, resting BP measured in office
Serum Assay: Lipid Profile | 8 weeks
  Total cholesterol, HDL-cholesterol, LDL-cholesterol, total triglycerides, ApoB, ApoA1, sdLDL, Lp(a)
Serum or Plasma Assay: Inflammatory Markers | 8 weeks
  MPO, LP-PLA2, hsCRP, ADMA/SDMA, oxLDL

OTHER OUTCOMES:
Number of subjects with abnormal haematology | 8 weeks
Number of subjects with abnormal clinical chemistry | 8 weeks
Number of subjects with abnormal kidney function | 8 weeks
Number of subjects with abnormal liver function | 8 weeks
Number of subjects with abnormal blood electrolytes | 8 weeks
Number of subjects with abnormal blood pressure | 8 weeks
Number of subjects with abnormal heart rate | 8 weeks
Incidence of Adverse Events | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (2):
- Canada (2):
  - KGK Synergize Inc., London, Ontario
  - Manna Research - Toronto, Toronto, Ontario